CLINICAL TRIAL: NCT07096063
Title: Comparative Effectiveness of Tirzepatide and Semaglutide in Individuals at Cardiovascular Risk
Acronym: TIRZSEMA-CVOT
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-TIRZSEMA-CVOT
Record Dates: First submitted 2025-07-23; First posted 2025-07-31 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes; Overweight; Cardiovascular (CV) Risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Tirzepatide; dulaglutide; semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: Tirzepatide vs dulaglutide
  Interventions: Drug: Tirzepatide; Drug: Dulaglutide
- Cohort 2: Semaglutide vs sitagliptin
  Interventions: Drug: Semaglutide; Drug: Sitagliptin
- Cohort 3: Tirzepatide vs semaglutide
  Interventions: Drug: Tirzepatide; Drug: Semaglutide

INTERVENTIONS:
Drug: Tirzepatide — New use of tirzepatide dispensing claim is used as the exposure.
  Groups: Cohort 1; Cohort 3
Drug: Dulaglutide — New use of dulaglutide dispensing claim is used as the comparator.
  Groups: Cohort 1
Drug: Semaglutide — New use of semaglutide dispensing claim is used as the exposure/comparator.
  Groups: Cohort 2; Cohort 3
Drug: Sitagliptin — New use of sitagliptin dispensing claim is used as the comparator.
  Groups: Cohort 2

SUMMARY:
Investigators are building an empirical evidence base for real-world data through large-scale emulation of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the Randomized Controlled Trials Duplicated Using Prospective Longitudinal Insurance Claims: Applying Techniques of Epidemiology (RCT-DUPLICATE) initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to assess the comparative effectiveness of

1. Tirzepatide vs dulaglutide,
2. Semaglutide vs sitagliptin,
3. Tirzepatide vs semaglutide

on cardiovascular outcomes in individuals typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes (T2DM) and overweight but might not meet the eligibility criteria of pivotal RCTs for each drug (SUSTAIN-6 and SURPASS-CVOT trials), used to support regulatory approval in patients at cardiovascular risk.Although many features of the target trials cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the target trial. Randomization cannot be achieved in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice.

The three database studies will be new-user active-comparative studies, conducted using 3 national United States claims databases, where investigators compare the effect of semaglutide vs sitagliptin (used as an active comparator placebo proxy), tirzepatide vs dulaglutide, and tirzepatide vs semaglutide on the composite end point of all-cause mortality, myocardial infarction, or stroke. Clinical guidelines during the study period recommended both tirzepatide and semaglutide for the same indications of glucose lowering and weight reduction.

ELIGIBILITY:
ELIGIBILITY FOR TIRZEPATIDE VS DULAGLUTIDE

Inclusion criteria

* History of MI, stroke, any surgical or percutaneous revascularization procedure, use of any antihypertensive/lipid-lowering drugs, coronary/carotid/peripheral artery disease, hypertension
* Type 2 diabetes
* BMI ≥25.0kg/m2
* Age ≥18 years
* Male or female sex

Exclusion Criteria:

* Medullary thyroid carcinoma, MEN syndrome type 2
* Malignancy
* Type 1 diabetes or secondary diabetes
* Chronic kidney disease or dialysis
* Uncontrolled diabetic retinopathy or maculopathy
* Pregnancy
* Prior use of pramlintide or any GLP-1-RA

ELIGIBILITY FOR SEMAGLUTIDE VS SITAGLIPTIN

Inclusion Criteria:

* History of MI, stroke, any surgical or percutaneous revascularization procedure, use of any antihypertensive/lipid-lowering drugs, coronary/carotid/peripheral artery disease, hypertension
* Type 2 diabetes
* BMI ≥25.0kg/m2
* Age ≥18 years
* Male or female sex

Exclusion Criteria:

* Medullary thyroid carcinoma, MEN syndrome type 2
* Malignancy
* Type 1 diabetes or secondary diabetes
* Chronic kidney disease or dialysis
* Uncontrolled diabetic retinopathy or maculopathy
* Pregnancy
* Prior use of pramlintide or any GLP-1-RA or DPP4i

ELIGIBILITY FOR TIRZEPATIDE VS SEMAGLUTIDE

Inclusion Criteria:

* History of MI, stroke, any surgical or percutaneous revascularization procedure, use of any antihypertensive/lipid-lowering drugs, coronary/carotid/peripheral artery disease, hypertension
* Type 2 diabetes
* BMI ≥25.0kg/m2
* Age ≥18 years
* Male or female sex

Exclusion Criteria:

* Medullary thyroid carcinoma, MEN syndrome type 2
* Malignancy
* Type 1 diabetes or secondary diabetes
* Chronic kidney disease or dialysis
* Uncontrolled diabetic retinopathy or maculopathy
* Pregnancy
* Prior use of pramlintide or any GLP-1-RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes mellitus and overweight.
Sampling Method: Non-Probability Sample
Enrollment: 887132 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, myocardial infarction or stroke (Tirzepatide vs. dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on the composite of all-cause mortality, myocardial infarction, or death in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Composite of all-cause mortality, myocardial infarction or stroke (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the composite of all-cause mortality, myocardial infarction, or death in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Composite of all-cause mortality, myocardial infarction or stroke (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs semaglutide on the composite of all-cause mortality, myocardial infarction, or death in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.

SECONDARY OUTCOMES:
Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring intravenous diuretics (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on all-cause mortality, hospitalization for heart failure, or urgent heart failure visits in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Urinary tract infections (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on the safety outcome of urinary tract infections in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Serious bacterial infections (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on the safety outcome of serious bacterial infections in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Gastrointestinal adverse events (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs dulaglutide on the safety outcome of gastrointestinal adverse events in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring intravenous diuretics (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of injectable semaglutide vs sitagliptin on all-cause mortality, hospitalization for heart failure, or urgent heart failure visits in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Urinary tract infections (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the safety outcome of urinary tract infections in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Serious bacterial infections (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the safety outcome of serious bacterial infections in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Gastrointestinal adverse events (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of injectable semaglutide vs sitagliptin on the safety outcome of gastrointestinal adverse events in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the individual components of the primary endpoint, i.e., all-cause mortality, myocardial infarction, or stroke in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Composite of all-cause mortality, hospitalization for heart failure, or urgent heart failure visits requiring intravenous diuretics (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs injectable semaglutide on all-cause mortality, hospitalization for heart failure, or urgent heart failure visits in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Urinary tract infections (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the safety outcome of urinary tract infections in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Serious bacterial infections (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the safety outcome of serious bacterial infections in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Gastrointestinal adverse events (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the comparative effect of tirzepatide vs injectable semaglutide on the safety outcome of gastrointestinal adverse events in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.

OTHER OUTCOMES:
Hernia (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs dulaglutide on negative control outcomes, including hernia in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Lumbar radiculopathy (Tirzepatide vs dulaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs dulaglutide on negative control outcomes, including lumbar radiculopathy in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Hernia (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of semaglutide vs sitagliptin on negative control outcomes, including hernia in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Lumbar radiculopathy (Injectable semaglutide vs sitagliptin) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of semaglutide vs sitagliptin on negative control outcomes, including lumbar radiculopathy in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Hernia (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs injectable semaglutide on negative control outcomes, including hernia, in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.
Lumbar radiculopathy (Tirzepatide vs injectable semaglutide) | 1 day after cohort entry date until the first of outcome or censoring, up to 365 days
  To evaluate the effect of tirzepatide vs injectable semaglutide on negative control outcomes, including lumbar radiculopathy, in patients typically treated in clinical practice who are at cardiovascular risk with type 2 diabetes and overweight.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital; Nils Krüger, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kruger N, Schneeweiss S, Desai RJ, Sreedhara SK, Kehoe AR, Fuse K, Hahn G, Schunkert H, Wang SV. Cardiovascular outcomes of semaglutide and tirzepatide for patients with type 2 diabetes in clinical practice. Nat Med. 2025 Nov 9. doi: 10.1038/s41591-025-04102-x. Online ahead of print. PMID 41207920

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT07096063/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Amendment to Study Protocol and Statistical Analysis Plan (2025-10-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT07096063/Prot_SAP_002.pdf